CLINICAL TRIAL: NCT04712331
Title: Effect of Preoperative Graduated Abdominal Exercises and Russian Stimulation on The Abdominal Muscles Strength After Abdominoplasty
Brief Title: Effect of Abdominal Exercises and Russian Stimulation on The Abdominal Muscles Strength After Abdominoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed E. Ali, Ph. D Candidate., Assistant Lecturer, South Valley University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002578
Record Dates: First submitted 2021-01-11; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Abdominoplasty
Keywords: abdominoplasty; Abdominal Exercises; Ultrasonography; Muscle Strength; Russian stimulation

STUDY DESIGN:
Intervention Model Description: Sixty patients will undergo abdominoplasty, their age ranged from 20 to 45 years, they were randomly distributed into four equal groups. The ultrasonography was used to evaluate abdominal muscle thickness as indicator for muscle strength at 4 occasions, initial assessment, pre-operative assessment, 2 months post-operative assessment, and finally 4 months post-operative assessment). For study group (A); received graduated abdominal exercises, group (B); received Russian stimulation on abdominal muscles, group (c); received combination between graduated abdominal exercises and Russian stimulation on abdominal muscles, the study groups received the treatment protocol for 30 min., 3 times per week for 6 weeks preoperatively for control group (D); were instructed to presume in normal activities of daily living preoperatively
Who Masked: Outcomes Assessor
Masking Description: Blinding process to participants and care providers was impossible due to the nature of intervention therapy. Data were analyzed by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: groups (A) & (B) & (C) ( three study groups ) and group (D) ( control group )
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The Study group A (Experimental): they received graduated abdominal strengthening exercises for 30 min., 3 times per week for 6 weeks preoperatively.
  Interventions: Other: Graduated abdominal strengthening exercises
- The Study group B (Experimental): they received Russian stimulation on abdominal muscles for 30 min., 3 times per week for 6 weeks preoperatively.
  Interventions: Device: The Russian current stimulation
- The Study group C (Experimental): they received combination between graduated abdominal strengthening exercises and Russian stimulation on abdominal muscles for 30 min., 3 times per week for 6 weeks preoperatively.
  Interventions: Other: Combination Product: Graduated abdominal strengthening exercises and the Russian current stimulation
- The Control group D (No Intervention): they were instructed to presume in normal activities of daily living preoperatively, without abdominal exercises or Russian stimulation.

INTERVENTIONS:
Other: Graduated abdominal strengthening exercises — Graduated abdominal strengthening exercises
  In this study the following equipments will be used to achieve treatment approaches:
  Exercise mat and inflatable Swiss ball 55 cm & 65 cm diameter. Wall bar, wedges, elastic tubing (Thera-band) with resistance ranges from light to very heavy (yellow, red, blue, green, and gray colors).
  Arms: The Study group A
Device: The Russian current stimulation — The Russian current is used for enhancing muscle; the muscular fiber by the electric stimulation.
  Arms: The Study group B
Other: Combination Product: Graduated abdominal strengthening exercises and the Russian current stimulation — Graduated abdominal strengthening exercises and the Russian current stimulation
  In this study the following equipments will be used to achieve treatment approaches:
  Exercise mat and inflatable Swiss ball 55 cm & 65 cm diameter. Wall bar, wedges, elastic tubing (Thera-band) with resistance ranges from light to very heavy (yellow, red, blue, green, and gray colors).
  The Russian current is used for enhancing muscle; the muscular fiber by the electric stimulation.
  Arms: The Study group C

SUMMARY:
To investigate the effect of preoperative graduated abdominal exercises and Russian stimulation on the abdominal muscles' strength after abdominoplasty

DETAILED DESCRIPTION:
To investigate the effect of preoperative graduated abdominal exercises and Russian stimulation on the abdominal muscles' strength after abdominoplasty. Sixty patients will undergo abdominoplasty, their age ranged from 20 to 45 years, they were randomly distributed into four equal groups. The ultrasonography was used to evaluate abdominal muscle thickness as indicator for muscle strength at 4 occasions, initial assessment, pre-operative assessment, 2 months post-operative assessment, and finally 4 months post-operative assessment). For study group (A); received graduated abdominal exercises, group (B); received Russian stimulation on abdominal muscles, group (c); received combination between graduated abdominal exercises and Russian stimulation on abdominal muscles, the study groups received the treatment protocol for 30 min., 3 times per week for 6 weeks preoperatively for control group (D); were instructed to presume in normal activities of daily living preoperatively

ELIGIBILITY:
Inclusion Criteria:

* Age range between 20-45 years. All patients desire an elective surgical repair.
* All patients were diagnosed with ventral hernia based on surgeon assessment.
* All patients will participate in the study.
* All patients enrolled to the study will have their informed consent.
* All patients are able to act in abdominal training program.
* All patients are able to follow orders during testing and training times.

Exclusion Criteria:

* A strangulated hernia.
* History of surgical interference (abdominal surgery) less than one year.
* Liver cirrhosis with or without ascites.
* Hip or spine deformities or contractures.
* Bowel obstruction, peritonitis, or perforation.
* Local or systemic infection.
* Patient is pregnant or intended to become pregnant during this period.
* Patient has indication for urgent surgery determinate by surgeon.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Abdominal muscles peak torque | first or initial assessment at day 0.
  Peak torque is the single highest torque output of the joint produced by muscular contraction as the limb moves through the range of motion.
Abdominal muscles peak torque | second or preoperative assessment after 42 days of treatment.
  Peak torque is the single highest torque output of the joint produced by muscular contraction as the limb moves through the range of motion.
Abdominal muscles peak torque | third assessment at 2 months post-operative.
  Peak torque is the single highest torque output of the joint produced by muscular contraction as the limb moves through the range of motion.
Abdominal muscles peak torque | fourth assessment at 4 months post-operative.
  Peak torque is the single highest torque output of the joint produced by muscular contraction as the limb moves through the range of motion.
Abdominal muscles thickness | first or initial assessment at day 0.
  it is a method for muscle strength measurement as muscle strength is correlated to its cross section or diameter.
Abdominal muscles thickness | second or preoperative assessment after 42 days of treatment.
  it is a method for muscle strength measurement as muscle strength is correlated to its cross section or diameter.
Abdominal muscles thickness | third assessment at 2 months post-operative.
  it is a method for muscle strength measurement as muscle strength is correlated to its cross section or diameter.
Abdominal muscles thickness | fourth assessment at 4 months post-operative.
  it is a method for muscle strength measurement as muscle strength is correlated to its cross section or diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed E. Ali, Ph.D student, Principal Investigator — South Valley University; Ayman M. Elmakaky, Principal Investigator — South Valley University
Locations (1):
- South Valley University, Faculty of Physical Therapy, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Vries CEE, Klassen AF, Hoogbergen MM, Alderman AK, Pusic AL. Measuring Outcomes in Cosmetic Abdominoplasty: The BODY-Q. Clin Plast Surg. 2020 Jul;47(3):429-436. doi: 10.1016/j.cps.2020.03.003. Epub 2020 Apr 17. PMID 32448479
- [Result] Le Roy B, Selvy M, Slim K. The concept of prehabilitation: What the surgeon needs to know? J Visc Surg. 2016 Apr;153(2):109-12. doi: 10.1016/j.jviscsurg.2016.01.001. Epub 2016 Feb 3. PMID 26851994
- [Result] Knight KA, Moug SJ, West MA. Systematic review: the impact of exercise on mesenteric blood flow and its implication for preoperative rehabilitation. Tech Coloproctol. 2017 Mar;21(3):185-201. doi: 10.1007/s10151-017-1589-9. Epub 2017 Feb 27. PMID 28243813
- [Result] Valkenet K, van de Port IG, Dronkers JJ, de Vries WR, Lindeman E, Backx FJ. The effects of preoperative exercise therapy on postoperative outcome: a systematic review. Clin Rehabil. 2011 Feb;25(2):99-111. doi: 10.1177/0269215510380830. Epub 2010 Nov 8. PMID 21059667
- [Result] Park SH, Hwangbo G. Effects of combined application of progressive resistance training and Russian electrical stimulation on quadriceps femoris muscle strength in elderly women with knee osteoarthritis. J Phys Ther Sci. 2015 Mar;27(3):729-31. doi: 10.1589/jpts.27.729. Epub 2015 Mar 31. PMID 25931718

DOCUMENTS (1):
  • Study Protocol (2021-01-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT04712331/Prot_000.pdf